CLINICAL TRIAL: NCT03533218
Title: A Novel Training Simulator for Portable Ultrasound Identification of Incorrect Newborn Endotracheal Tube Placement, Karachi Pakistan
Brief Title: A Novel Training Simulator for Portable Ultrasound Identification of Incorrect Newborn Endotracheal Tube Placement
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: The Hospital for Sick Children (Other); Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Dr Shabina Ariff, Associate Professor, Aga Khan University
Other Study IDs: POCUS
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Point of Care Ultrasound
Keywords: endotracheal tube, point of care ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Point of care Ultrasound machine — POCUS methods of assessing ETT location offer an alternative that is time saving and thereby of critical importance in the neonatal "time-is-brain" scenario. Recently the government of Pakistan began upgrading health facilities and ensuring placement of essential equipment required to provide competent medical care, which may include provision of ultrasound machines to areas where there is established benefits to their use. Presence of trained staff and provision of portable ultrasound machine with short start-up time can save newborn lives(12).POCUS method empowers health care providers to read and interpret images in real time thereby saving critical time and need for specialized human resources (radiologists).

SUMMARY:
First seconds after birth, new born baby go through physiologic changes to successfully adjust to the external environment specially establishment of independent respiration. Majority of the organ systems adaptation in newborns occur gradually, but radical and rapid cardiopulmonary adaptation must occur for neonates to survive. It is during this period that approximately 10% neonates require some level of support in the form of resuscitation.

A knowledgeable, quick and skillful response by all caregivers is crucial for extra uterine survival. Tracheal intubation is performed frequently in the Neonatal Intensive Care Units (NICU) and delivery rooms. Neonatal intubation is a critical and time-sensitive procedure, and failure deprives the sickest newborns of oxygen.

Current methods to detect a misplaced esophageal ETT in newborns are suboptimal. Physical examination findings are often unreliable, exhaled carbon-dioxide testing is often unavailable outside of resource-rich facilities and can lead to false positive results ,while chest radiographs are not only time consuming ,labor intensive but also expose vulnerable newborn babies to significant radiation However portable ultrasound machines are relatively available even in small centers mostly being used in the maternity units, being an indispensable tool for managing obstetrics, gynecology and trauma cases.

POCUS methods of assessing ETT position offer an alternative that is time saving, cheap and safe, thereby of critical importance in the neonatal "time-is-brain" scenario.

Our project aims to demonstrate that POCUS can effectively and accurately detect esophageal intubations, and in shorter period of time than current standard-of-care methods that are colorimetric end- tidal carbon-dioxide (CO2) detector and chest x-ray.

DETAILED DESCRIPTION:
Phase 1 would entirely base on training of all newborn care providers. The training phase of the study includes two stages:

Stage 1: It will involve training of new born care providers in detecting esophageal versus tracheal intubations using the ultrasound simulator, and then ensure they are able to accurately detect this difference using our evaluation tools.

Experts in POCUS will train neonatal health care providers at Aku.

Stage 2 : It would comprise of validation and assessment of POCUS competency. For this purpose neonatal health care providers that underwent training will perform Ultrasound of intubated babies who are hemodynamically stable in NICU, captured images and save them.

These images will be interpreted in real time by the trainee and validate by trained PI. 10% images will be sent to Sick Kids POCUS trainer for revalidation. Health care provider will validate at least 10 images correctly to be certified as successfully trained and move to Phase 2.

Phase 2. New-born at The Aga Khan Hospital who requires intubation will be assessed for ETT placement via ultrasound and simultaneously with the standard methods. The time required to assess a correct endotracheal intubation will be compared between POCUS and standard care methods that are colorimetric end- tidal carbon-dioxide (CO2) detector.

Study population and sample size:

Phase 1: The training session will be provided to health care providers who attend deliveries and exclusively involved in newborn care, which include Neonatal attending, postgraduate trainees, neonatal fellows and nursing staffs.

The POCUS will be done by Fellows, attending and Senior Staff only.

Phase 2: A Sample size of 292 newborn will be recruited considering these assumptions that in the Aga khan university, Hospital Karachi currently has approximately 5,000 deliveries per year and 600 infants per year require admission in the NICU (12% of total NICU admissions).

ELIGIBILITY:
phase I

Inclusion Criteria All healthcare workers who are involved in assessing ETT location in newborns after intubation using standard methods at AKUH

Exclusion Criteria

-Providers who are not involved in newborn resuscitation and assessing ETT location using standard methods

phase II Inclusion Criteria - All newborns needing intubation in the delivery room or in the NICU

Exclusion Criteria

- Newborns with any congenital syndromes affecting the oropharynx or airway anatomy.

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: phase I health care workers who currently perform standard-of-care ETT location assessment in the delivery room or NICU.
  phase II all newborns require intubation in labor and delivery room or in NICU.
Sampling Method: Probability Sample
Enrollment: 292 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
training of health care workers | 4 months
  To determine if neonatal providers trained in ETT location with the simulator will detect correct ETT placement with >95% accuracy immediately and after validation of their skills.

SECONDARY OUTCOMES:
comparison with standard methods | 12 months
  To determine the time to detect ETT location is less for POCUS than for colorimetric end- tidal carbon-dioxide (CO2) detector and chest radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Shabina Ariff, MBBS, FCPS, Principal Investigator — Aga Khan University; Mark Tessaro, MD, FRCPC, Study Chair — The Hospital for Sick Kids; Khushboo Qaim, BScN, Study Director — Aga Khan University; Hasan Meerali, MD, FAAP, Study Director — The Hospital for Sick Kids
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Askin DF. Complications in the transition from fetal to neonatal life. J Obstet Gynecol Neonatal Nurs. 2002 May-Jun;31(3):318-27. doi: 10.1111/j.1552-6909.2002.tb00054.x. PMID 12033545
- [Background] Simpson K, & Chreehan, P. Newborn adaptation to extrauterine life. Perinatal nursing,. 2nd ed. ed. PA7 Lippincott: Philadelphia; (2001).
- [Background] Stenson BJ, Boyle DW, Szyld EG. Initial ventilation strategies during newborn resuscitation. Clin Perinatol. 2006 Mar;33(1):65-82, vi-vii. doi: 10.1016/j.clp.2005.11.015. PMID 16533634
- [Background] American Academy of Pediatrics/American Heart Association. American Academy of Pediatrics/American Heart Association clarification of statement on cardiovascular evaluation and monitoring of children and adolescents with heart disease receiving medications for ADHD: May 16, 2008. J Dev Behav Pediatr. 2008 Aug;29(4):335. doi: 10.1097/DBP.0b013e31318185dc14. No abstract available. PMID 18698199
- [Background] Schmolzer GM, Kumar M, Pichler G, Aziz K, O'Reilly M, Cheung PY. Non-invasive versus invasive respiratory support in preterm infants at birth: systematic review and meta-analysis. BMJ. 2013 Oct 17;347:f5980. doi: 10.1136/bmj.f5980. PMID 24136633
- [Background] Jukkala AM, Henly SJ. Readiness for neonatal resuscitation: measuring knowledge, experience, and comfort level. Appl Nurs Res. 2007 May;20(2):78-85. doi: 10.1016/j.apnr.2006.01.006. PMID 17481471
- [Background] Carbajal R, Eble B, Anand KJ. Premedication for tracheal intubation in neonates: confusion or controversy? Semin Perinatol. 2007 Oct;31(5):309-17. doi: 10.1053/j.semperi.2007.07.006. PMID 17905186
- [Background] Schmolzer GM, O'Reilly M, Davis PG, Cheung PY, Roehr CC. Confirmation of correct tracheal tube placement in newborn infants. Resuscitation. 2013 Jun;84(6):731-7. doi: 10.1016/j.resuscitation.2012.11.028. Epub 2012 Dec 1. PMID 23211476
- [Background] Peterson J, Johnson N, Deakins K, Wilson-Costello D, Jelovsek JE, Chatburn R. Accuracy of the 7-8-9 Rule for endotracheal tube placement in the neonate. J Perinatol. 2006 Jun;26(6):333-6. doi: 10.1038/sj.jp.7211503. PMID 16642028
- [Background] Divatia J, Bhowmick K. Complications of endotracheal intubation and other airway management procedures. Indian J Anaesth. 2005;49(4):308-18.
- [Background] Adi O, Chuan TW, Rishya M. A feasibility study on bedside upper airway ultrasonography compared to waveform capnography for verifying endotracheal tube location after intubation. Crit Ultrasound J. 2013 Jul 4;5(1):7. doi: 10.1186/2036-7902-5-7. PMID 23826756
- [Background] Sakhuja P, Finelli M, Hawes J, Whyte H. Is It Time to Review Guidelines for ETT Positioning in the NICU? SCEPTIC-Survey of Challenges Encountered in Placement of Endotracheal Tubes in Canadian NICUs. Int J Pediatr. 2016;2016:7283179. doi: 10.1155/2016/7283179. Epub 2016 Jan 19. PMID 26884771
- [Background] Demographic P. Health Survey 2012-13: Islamabad. Pakistan, and Calverton, Maryland USA: National Institute of Population Studies and ICF International. 2013.
- [Background] Jehan I, Harris H, Salat S, Zeb A, Mobeen N, Pasha O, McClure EM, Moore J, Wright LL, Goldenberg RL. Neonatal mortality, risk factors and causes: a prospective population-based cohort study in urban Pakistan. Bull World Health Organ. 2009 Feb;87(2):130-8. doi: 10.2471/blt.08.050963. PMID 19274365
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Aga Khan University From Wikipedia, the free encyclopedia [07.03.2017].
- [Background] Chou EH, Dickman E, Tsou PY, Tessaro M, Tsai YM, Ma MH, Lee CC, Marshall J. Ultrasonography for confirmation of endotracheal tube placement: a systematic review and meta-analysis. Resuscitation. 2015 May;90:97-103. doi: 10.1016/j.resuscitation.2015.02.013. Epub 2015 Feb 21. PMID 25711517
- [Derived] Ali KQ, Soofi SB, Hussain AS, Ansari U, Morris S, Tessaro MO, Ariff S, Merali H. Simulator-based ultrasound training for identification of endotracheal tube placement in a neonatal intensive care unit using point of care ultrasound. BMC Med Educ. 2020 Nov 7;20(1):409. doi: 10.1186/s12909-020-02338-4. PMID 33160342
- [Derived] Merali HS, Tessaro MO, Ali KQ, Morris SK, Soofi SB, Ariff S. A novel training simulator for portable ultrasound identification of incorrect newborn endotracheal tube placement - observational diagnostic accuracy study protocol. BMC Pediatr. 2019 Nov 13;19(1):434. doi: 10.1186/s12887-019-1717-y. PMID 31722685